CLINICAL TRIAL: NCT02306265
Title: Assessment of Diagnostic Accuracy and Performance of Digital Breast Tomosynthesis Compared to Mammography (ADAPT Trial) ADAPT-SCR: Recruitment Plan for Asymptomatic Women Undergoing Screening Mammography
Brief Title: Assessment of Diagnostic Accuracy and Performance of Digital Breast Tomosynthesis Compared to Mammography
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 124.03-2014-GES-0010
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Tumors, Breast; Cancer Screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBT and FFDM (Other): Subjects will undergo 2D breast imaging with full-field digital mammography (FFDM) device (active comparator) and 3D breast imaging with digital breast tomosynthesis (DBT) device (experimental).
  Interventions: Device: FFDM; Device: DBT

INTERVENTIONS:
Device: FFDM — 2D imaging of the breast using Full-Field Digital Mammography (FFDM) device
  Other Names: Full-Field Digital Mammogram; 2D breast imaging
Device: DBT — 3D imaging of the breast using Digital Breast Tomosynthesis (DBT) device
  Other Names: Digital Breast Tomosynthesis; 3D breast imaging

SUMMARY:
The aim of this recruitment plan (ADAPT-SCR) is to collect image and other data on both digital breast tomosynthesis (DBT) and full-field digital mammography (FFDM) from asymptomatic women undergoing screening mammography.

DETAILED DESCRIPTION:
ADAPT program consists of 2 recruitment plans (ADAPT-SCR and ADAPT-BX) followed by an off-line read of the images and data collected (ADAPT-BIE). This study involves the comparison of two devices that can identify abnormalities in routine breast screening and diagnostic mammography. Mammography is usually done with full-field digital mammography (FFDM), which takes flat, two-dimensional X-ray images of the breast. Doctors use the two-dimensional images to look for cancers and other abnormal tissue. The purpose of this study is to learn more about the accuracy of full-field digital mammography devices and a new mammography device called digital breast tomosynthesis (DBT). DBT is similar to full-field digital mammography, but can also move around the breast to get X-ray images from different angles, which provides a three-dimensional view that doctors can use to look for cancers and abnormal tissue. Subjects will undergo routine imaging with FFDM and will also have a DBT performed. They will continue with their standard of care treatment as would occur outside of the study. Based on the results of the FFDM and DBT, the subject's status will be followed-up with routing imaging at approximately 1 year (10-16 months). If the doctor recommends biopsy based on the FFDM or DBT, information about the biopsy and cancer determination results will be collected. Being in this study does not require subjects to have a biopsy that was not recommended by the doctor for normal medical care.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 years or older (≥30 years old);
* Asymptomatic women scheduled for screening mammography or have completed a screening mammogram within the past 30 days;
* Mammography completed on a General Electric (GE) GE FFDM system (with craniocaudal (CC) and mediolateral oblique (MLO) views) at the site or another clinical facility;
* Are able and willing to comply with study procedures;
* Have signed and dated the informed consent form;
* Are either surgically sterile or postmenopausal or, if of childbearing potential, the possibility of pregnancy is remote based on a documented negative patient history and, optionally, a negative urine pregnancy test (if subject requests one).

Exclusion Criteria:

* Have been previously included in this study;
* Have a history of breast cancer and are in active treatment. However, subjects with a prior lumpectomy (> 5 years prior) who receive only routine screening mammography views can be included;
* Have breasts too large to be adequately positioned on 24 x 31 centimeter (cm) FFDM digital receptor without anatomical cut off during either FFDM or DBT examination;
* Have participated in (within the prior 30 days) another trial of an investigational product expected to interfere with study procedures or outcomes;
* Have breast implant(s);
* Have reconstructed breast(s).

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray Rebner, MD, Principal Investigator — Beaumont Health; William Poller, MD, Principal Investigator — West Penn Allegheny Health System
Locations (2):
- United States (2):
  - Beaumont Health System, Royal Oak, Michigan
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject population consisted of asymptomatic adult women (30 years of age or greater) scheduled for routine screening mammography.
Groups:
- Mammography FFDM and DBT: All subjects were expected to undergo 2D breast imaging with full-field digital mammography (FFDM) and 3D breast imaging with digital breast tomosynthesis (DBT). The order in which these scans took place was not assigned.
  Digital Breast Tomosynthesis: 3D imaging of the breast using Digital Breast Tomosynthesis (DBT) device
  Full-Field Digital Mammogram: 2D imaging of the breast using Full-Field Digital Mammography (FFDM) device
Period: Overall Study
Arm/Group | Mammography FFDM and DBT
Started | 250
Completed | 249
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of asymptomatic adult women (>30 years of age) scheduled for routine screening mammography. All women followed the same participant flow plan, and were all considered to be in the same single arm of the study.
Groups:
- Mammography FFDM and DBT: All subjects underwent 2D breast imaging with full-field digital mammography (FFDM) followed by 3D breast imaging with digital breast tomosynthesis (DBT). Order for scan method was not assigned.
  Digital Breast Tomosynthesis: 3D imaging of the breast using Digital Breast Tomosynthesis (DBT) device
  Full-Field Digital Mammogram: 2D imaging of the breast using Full-Field Digital Mammography (FFDM) device
Arm/Group | Mammography FFDM and DBT
Number analyzed (Participants) | 250
Age, Continuous [Mean (Full Range); unit: years] | 57.4 [39 to 83]
Sex: Female, Male [Count of Participants; unit: Participants] — Per Inclusion/Exclusion criteria, all study participants were female
  Participants
    Female | 250
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 250
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 250
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 250
Successfully completed FFDM and DBT scans [Count of Participants; unit: Participants] — This baseline measure includes enrolled participants who successfully completed both DBT and FFDM scans.
  Participants | 249

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Imaging Data Collected
Description: Collect breast image data using two (2) methods: Digital Breast Tomosynthesis (DBT) and Full Field Digital Mammography (FFDM) from asymptomatic women undergoing screening mammography.
Time Frame: within 30 days of enrollment
Population: The efficacy population for primary outcome were subjects meeting study inclusion/exclusion criteria with no protocol violations judged to affect the ability to evaluate the subject, whose DBT/FFDM images were diagnostically evaluable and whose mammography images were available for independent blinded evaluation, regardless of image quality.
Measure: Count of Participants; unit: Participants
Groups:
- Mammography FFDM and DBT: Subjects underwent 2D breast imaging with full-field digital mammography (FFDM) followed by 3D breast imaging with digital breast tomosynthesis (DBT).
  Digital Breast Tomosynthesis: 3D imaging of the breast using Digital Breast Tomosynthesis (DBT) device
  Full-Field Digital Mammogram: 2D imaging of the breast using Full-Field Digital Mammography (FFDM) device
Arm/Group | Mammography FFDM and DBT
Number analyzed (Participants) | 250
Participants
  Participants with images collected by both methods | 249
  Participants with image collected by one method | 1

2. Other Pre Specified Outcome: Device Malfunctions by Modality (DBT or FFDM).
Description: Number of device malfunctions by modality (DBT or FFDM)
Time Frame: Duration of study -approximately 26 months
Population: One device malfunction reported for FFDM; Zero device malfunctions reported for DBT.
Measure: Number; unit: Malfunctions
Groups:
- Mammography FFDM and DBT: All subjects underwent 2D breast imaging with full-field digital mammography (FFDM) and 3D breast imaging with digital breast tomosynthesis (DBT). The order in which these scans took place was not assigned.
  Digital Breast Tomosynthesis: 3D imaging of the breast using Digital Breast Tomosynthesis (DBT) device
  Full-Field Digital Mammogram: 2D imaging of the breast using Full-Field Digital Mammography (FFDM) device
Arm/Group | Mammography FFDM and DBT
Number analyzed (Participants) | 250
Malfunctions
  Device malfunctions reported for FFDM | 1
  Device malfunctions reported for DBT | 0

3. Other Pre Specified Outcome: Cancer-positive Participants
Description: Participants confirmed to be positive for cancer on histology review.
Time Frame: Duration of study - approximately 26 months
Population: Participants who completed the study, including conclusive histology review, and cancer status was positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Mammography FFDM and DBT
Number analyzed (Participants) | 188
Participants | 6

ADVERSE EVENTS:
Time Frame: Time frame in which subjects were to complete the two scan types (up to 30 days).
Description: Adverse Event (AE): As defined by European Norms International Standard Organization (EN ISO) ISO 14155-2011: any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.
Arm/Group | Mammography FFDM and DBT
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 2/250
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mammography FFDM and DBT (N=250)
Rash (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
The aim of this study (ADAPT-SCR) was to collect image data using two methods from asymptomatic women undergoing screening mammography. No statistical hypothesis was tested in this image collection study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT02306265/Prot_SAP_000.pdf